CLINICAL TRIAL: NCT03127124
Title: An Open-label, Multicenter, Single-arm, Phase 1b/2 Study of NANT-008 in Combination With 5-fluorouracil, Bevacizumab, Leucovorin, and Oxaliplatin in Patients With Metastatic Pancreatic Adenocarcinoma.
Brief Title: QUILT-2.022 NANT-008 in Combination w/ 5-fluorouracil, Bevacizumab, Leucovorin & Oxaliplatin in Subjects With Pancreatic Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was withdrawn due to no enrollment
Sponsor: NantPharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-2.022
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2020-06

CONDITIONS: Pancreatic Adenocarcinoma Metastatic
MeSH Terms: interventions — Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NANT-008 in combination with other agents (Experimental): NANT-008 will be administered in combination with 5-fluorouracil, bevacizumab, leucovorin, and oxaliplatin in patients with metastatic pancreatic adenocarcinoma.
  Interventions: Drug: NANT-008; Drug: Fluorouracil Injectable Product; Drug: Avastin Injectable Product; Drug: Leucovorin Calcium Injection; Drug: Eloxatin Injectable Product

INTERVENTIONS:
Drug: NANT-008 — Paclitaxel: benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI)
Drug: Fluorouracil Injectable Product — 5-fluoro-2,4 (1H,3H)-pyrimidinedione.
Drug: Avastin Injectable Product — Recombinant humanized monoclonal IgG1 antibody
Drug: Leucovorin Calcium Injection — Calcium N -[p -[[[(6RS )-2-amino-5-formyl-5,6,7,8-tetrahydro-4-hydroxy-6-pteridinyl]methyl]amino]benzoyl]-L-glutamate (1:1).
Drug: Eloxatin Injectable Product — cis-[(1 R,2 R)-1,2-cyclohexanediamine-N,N'] [oxalato(2-)- O,O'] platinum.

SUMMARY:
This is a phase 1b/2 study to evaluate the safety and efficacy of NANT-008 in combination with 5-fluorouracil, bevacizumab, leucovorin, and oxaliplatin in patients with metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Phase 1b is designed to evaluate the recommended phase 2 dose (RP2D) of NANT-008 and dose-limiting toxicities (DLTs) of NANT-008 in combination with metronomic 5-FU, bevacizumab, leucovorin, and oxaliplatin in subjects with advanced metastatic pancreatic carcinoma. In phase 2, subjects will receive the combination of RP2D of NANT-008 from phase 1b in combination with metronomic 5-FU, bevacizumab, leucovorin, and oxaliplatin. Phase 2 is designed to evaluate the efficacy of the tested regimen as assessed by 1-year survival rate in subjects with advanced metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject is between ≥ 18 and ≤ 65 years of age at the time of signing the informed consent form (ICF).
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or IEC guidelines.
3. Histologically confirmed, unresectable, locally advanced or metastatic pancreatic adenocarcinoma.
4. ECOG performance status of 0 to 1.
5. Have at least 1 measurable lesion and/or non-measurable disease evaluable according to RECIST Version 1.1.
6. Have not received any prior treatment other than radiation therapy for symptomatic pain relief.
7. Resolution of all toxic side effects of prior chemotherapy, radiotherapy, or surgical procedures to CTCAE grade ≤ 1, with the exception of alopecia.
8. Must be willing to provide pre- and post-treatment blood samples for exploratory analyses.
9. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
10. Must have a recent FFPE tumor biopsy specimen following the conclusion of the most recent anticancer treatment and be willing to release the specimen for tumor molecular profiling analysis. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period.
11. Agreement to practice effective contraception (both male and female subjects, if the risk of conception exists).
12. Must have a stable, functioning stent at least 2 weeks before the beginning of the study (metal stents are preferred as per NCCN guidelines) if subject has had a previous biliary or pancreatic duct obstruction requiring stent placement.

Exclusion Criteria:

1. History of previous systemic chemotherapy or investigational therapy.
2. History of other active malignancies or brain metastasis except: controlled basal cell carcinoma or squamous cell carcinoma; prior history of in situ cancer (eg, breast, melanoma, squamous cell carcinoma of the skin, cervical) and > 5 years without evidence of disease; prior history of prostate cancer that is not under active systemic treatment (except hormonal therapy) and with undetectable PSA (< 0.2 ng/mL).
3. Inadequate organ function, evidenced by the following laboratory results:

   1. White blood cell (WBC) count < 3,500 cells/mm3
   2. Absolute neutrophil count < 1,500 cells/mm3.
   3. Platelet count < 100,000 cells/mm3.
   4. Hemoglobin < 9 g/dL.
   5. Total bilirubin greater than the upper limit of normal (ULN) at time of enrollment; unless the subject has known history of Gilbert's syndrome.
   6. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   7. Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   8. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   9. International normalized ratio (INR) or activated partial thromboplastin time (aPTT) or partial thromboplastin time (PTT) >1.5 × ULN.
4. Pre-existing peripheral neuropathy > grade 1 based on NCI CTCAE V4.03.
5. Dihydropyrimidine dehydrogenase gene polymorphism (DPYD*2A) (must be tested prior to inclusion).
6. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
7. Positive results of screening test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
8. Undergone major surgery, other than diagnostic surgery (ie, surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to day 1 of treatment in this study or surgical wound has not fully healed.
9. History of connective tissue disorders (eg, lupus, scleroderma, arteritis nodosa).
10. Evidence of gastric ulcers, gastrointestinal fistulas, and gastrointestinal perforations.
11. History of interstitial lung disease, history of slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies that in the opinion of the Investigator may put them at increased risk of interstitial pneumonitis.
12. Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication.
13. Recent history of clinically significant hemoptysis.
14. Known hypersensitivity to any component of the study medication(s).
15. Pregnant and nursing women.
16. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.
17. Concurrent or prior use of a strong CYP3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
18. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Phase 1b Primary Endpoint | 12 weeks
  Determine the recommended phase 2 dose (RP2D) of NANT-008 and dose-limiting toxicities (DLTs) of NANT-008
Phase 2 Primary Endpoint | 1 year
  Evaluate the efficacy of the tested regimen as assessed by the 1 year survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institutes for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: No